CLINICAL TRIAL: NCT00472914
Title: Initial Assessment of the Use of Surface Electromyography as a Tool for Clinical Evaluation of Hypertonia in Children
Brief Title: Use of EMG to Assess Clinical Hypertonia
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Other Study IDs: EMG auditory
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Cerebral Palsy; Hypertonia; Spasticity; Dystonia; Rigidity
Keywords: Hypertonia; Childhood
MeSH Terms: conditions — Cerebral Palsy; Muscle Hypertonia; Muscle Spasticity; Dystonia; Muscle Rigidity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: portable surface electromyography

SUMMARY:
A handheld surface electromyography device will be tested by clinicians on children with limb hypertonia, and inter-rater reliability will be assessed with and without the device.

DETAILED DESCRIPTION:
Hypothesis:

Qualitative surface EMG measurement during passive movement will increase the inter-rater reliability of clinicians for diagnosis of spasticity and dystonia in children with hypertonia.

Specific Aims:

1. Develop a handheld surface EMG device with auditory output that can be used similarly to a stethoscope to listen non-invasively to the activity of muscles.
2. Provide clinicians at 5 different institutions with a device to test for 2 months in their own clinics.
3. Bring all 5 clinicians to Stanford University for a single-day exercise in which each clinician will examine 10 children with hypertonia. Each clinician will rate the children without using the device, and then again with the device. Intra-class correlations and kappa statistics will be used to assess whether the use of the device leads to improved inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18
* hypertonia in at least one limb due to spasticity

Exclusion Criteria:

* any condition that would increase the risk of participation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence D Sanger, Md, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States